CLINICAL TRIAL: NCT03555864
Title: Peripheral Intravenous Cannulation With Support of Infrared Laser Vein Viewing System in Obese Patients
Brief Title: Intravenous Access Using Infrared Laser
Acronym: AccuV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, Clinical Professor, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: Local-PC-2017-2
Record Dates: First submitted 2017-12-30; First posted 2018-06-14 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Morbid; Obstetric Anesthesia Problems
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese: Patients need two intravenous access with infra red
  Interventions: Device: infrared transluminescent device

INTERVENTIONS:
Device: infrared transluminescent device — use of infra red for venous access for second intravenous access

SUMMARY:
Peripheral venous access is a prerequisite for anesthesiological for surgical patients.It is often difficult to establish and potentially painful in obese patients (Body mass Index > 35). AV300 uses near infrared laser light to improve visibility of peripheral veins and could help cannulating them. The aim of this study was to examine if use of Accuvein(®) AV300 vein viewer could facilitate venous cannulation in obese patients (surgical and obstetric).

ELIGIBILITY:
Inclusion Criteria

* > 18 years
* surgery that need double intravenous perfusion

Exclusion Criteria:

* < 18 years
* body mass index< 35
* refusal
* minor surgery that need only one intravenous access

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that need second intravenous access for surgery or obstetric
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
success for second intravenous line using infra red | 1 day
  number of attempts

SECONDARY OUTCOMES:
time | 1 day
  time in second for second intravenous access

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves Lefrant, MD,PhD, Study Chair — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU Nimes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No